CLINICAL TRIAL: NCT04692584
Title: Effects of Mother-Sung Lullabies on Vaccination-Induced Infant Pain and Maternal Anxiety
Brief Title: Effects of Mother-Sung Lullabies on Infant Pain and Maternal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Pınar BEKAR, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mehmet Akif Ersoy University
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-02

CONDITIONS: Pain; Anxiety
Keywords: Anxiety; Pain; Vaccination; Mother; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This was an experimental, randomized controlled study. These babies were randomly assigned to one of two groups, including 30 babies in the lullaby group and 30 babies in the control group. Randomization was performed using a sealed envelope method. The video recordings were evaluated by two academicians in the field of child health and disease nursing, including a researcher and a research assistant with a doctorate in child health and disease nursing who were not blinded to the group assignment. These observers were blinded to the other's observations and did not discuss the scores.
Masking Description: The video recordings were evaluated by two academicians in the field of child health and disease nursing, including a researcher and a research assistant with a doctorate in child health and disease nursing who were not blinded to the group assignment. For each assessment, the observers watched the videos of the babies and conducted NIPS assessments during and after the intervention. These observers were blinded to the other's observations and did not discuss the scores.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Lullaby Group (Experimental): In this group, their mothers sang a lullaby during the vaccination process. Each mother touched her baby's hands and body while singing a lullaby and hugged her baby after the procedure.
  Interventions: Behavioral: The Lullaby Group
- Control Group (No Intervention): In this group, their mothers did not sing a lullaby during the vaccination process.
  Mothers touched their infant's hands and body and talk to their infants during and after vaccination. Mothers hugged their infant after the procedure.

INTERVENTIONS:
Behavioral: The Lullaby Group — Approximately 15 seconds before the vaccination, each baby's mother began to sing a lullaby. Infant's mother continued to sing lullabies until all the vaccinations, which were given immediately after the BCG vaccination, were completed. Each mother touched her baby's hands and body while singing a lullaby and hugged her baby after the procedure. All the mothers sang the same lullaby, "Sleep and Grow". Mothers were reminded of the words to the lullaby before vaccine administration.
  Arms: The Lullaby Group

SUMMARY:
Childhood pain can cause long-term and psychologically harmful effects. Music can reduce pain and anxiety. This study aimed to investigate the effects of the mother-sung lullaby during vaccine administration on vaccine-induced pain in babies and anxiety in mothers.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of the mother-sung lullaby during vaccine administration on vaccine-induced pain in babies and anxiety in mothers. Two family health centers in Turkey between March 4, 2020, and August 28, 2020. A total of 60 babies who received the Bacille Calmette-Guérin vaccine and their mothers.These babies were randomly assigned to one of two groups, including 30 babies in the lullaby group and 30 babies in the control group. Data on descriptive information for all babies and mothers were collected through face-to-face interviews with the mothers before vaccination. Heart rate, oxygen saturation, and crying duration were measured in all babies. Heart rate and oxygen saturation of the babies were recorded using a pulse oximeter during and after vaccine administration. The crying time, measured for up to 30 seconds after vaccination, was recorded as the total cry time (using video seconds). The pain score was evaluated by two observers using the Neonatal Infant Pain Scale, based on video recordings obtained during and after vaccine administration. In addition, mothers' anxiety scores were measured using the "State Anxiety Inventory," both before and after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* gestational age of 37-42 weeks
* postnatal age at full two month
* receiving the Bacille Calmette-Guérin vaccine
* birth weight of 2500 gr or higher
* no congenital anomalies
* stable general condition
* not taking any pain medication before vaccination
* mothers were required to be older than 18 years and agree to participate in the study

Exclusion Criteria:

* taking analgesic medication within 4 hours before the procedure
* parents not willing to participate in research.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 6 MONTHS
  Neonatal Infant Pain Scale (NIPS) was used for the pain assessment. The NIPS consists of 6 behavioral sections, including facial expression, crying, breathing pattern, arm and leg movements, and wakefulness. Although 2 point values (0-1 point) can be scored for behaviors other than crying, 3 point values (0-1-2 points) are scored for crying. The total score ranges from 0 to 7, with higher scores indicated increased pain intensity.
State Anxiety Inventory (SAI) | 6 MONTHS
  The SAI was used in this study, which can be used to determines how an individual feels at a certain time and under certain conditions. The SAI consists of 20 questions, with scores ranging from 20-80. A high score indicates high anxiety, whereas a low score indicates low anxiety. The State Anxiety Inventory was used to determine the anxiety levels of the mothers before and after the vaccine administration.

SECONDARY OUTCOMES:
Heart Rate | 6 MONTHS
  Heart rate of the babies were recorded using a pulse oximeter placed on the right or left foot or hand of each baby before the intervention. Heart rate levels were recorded during and after vaccination.
Oxygen Saturation | 6 MONTHS
  Oxygen saturation of the babies were recorded using a pulse oximeter placed on the right or left foot or hand of each baby before the intervention. Oxygen saturation levels were recorded during and after vaccination.
Crying duration of babies | 6 MONTHS
  The crying time was expressed in seconds. The cry time measured up to 30 seconds after vaccination was the total cry time (using video seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Prof.Dr., Study Director — Akdeniz University, Department of Child Health and Disease Nursing
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bekar P, Efe E. Effects of mother-sung lullabies on vaccination-induced infant pain and maternal anxiety: A randomized controlled trial. J Pediatr Nurs. 2022 Jul-Aug;65:e80-e86. doi: 10.1016/j.pedn.2022.03.003. Epub 2022 Mar 25. PMID 35341657